CLINICAL TRIAL: NCT04533061
Title: Lung Transplant Patients' T Cell Responses to Influenza Vaccine Viruses Between Seasons
Brief Title: Influenza Vaccine in Lung Transplant Patients - T Cells
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: H-2004-0240a; A561000 (Other: UW Madison); PHARM/PHARMACY/PHARMACY (Other: UW Madison)
Record Dates: First submitted 2020-08-25; First posted 2020-08-31 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Influenza
Keywords: Lung transplant; Healthy
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lung Transplant, Vaccine: Cohort consist of individuals who have received lung transplants Inactivated influenza vaccine will be administered intramuscularly annually.
  Interventions: Drug: Influenza vaccine
- Healthy Control, Vaccine: Cohort consists of healthy individuals who received the influenza vaccine Inactivated influenza vaccine will be administered intramuscularly annually.
  Interventions: Drug: Influenza vaccine

INTERVENTIONS:
Drug: Influenza vaccine — influenza vaccine 0.5 ml intramuscularly each season
  2004-2005 season contains: A/New Caledonia/20/99 (H1N1)-like, A/Fujian/411/2002 (H3N2-like), and B/Shanghai/361/2002-like antigens
  2005-2006 season contains: A/New Caledonia/20/99 (H1N1)-like, A/California/7/2004 (H3N2), and B/Shanghai/361/2002-like antigens

SUMMARY:
This a sub-study of a 5-year study designed to investigate how antibody and T cell responses following influenza vaccine compare among lung transplant patients, patients waiting for lung transplantation, and healthy individuals.

This trial is designed to investigate the hypothesis that there is no difference in T Cell response to the influenza vaccine between lung transplant patients and healthy controls.

DETAILED DESCRIPTION:
Influenza virus infection causes significant morbidity and mortality each season. The infection is particularly serious in the elderly and those with chronic cardiopulmonary conditions. Solid organ transplant recipients receiving immunosuppressive therapy may be at particularly high risk for serious influenza infection. Lung transplant patients may have an even higher risk because of their underlying pathophysiology.

Influenza prophylaxis is extremely important in the care of the transplant patient. Annual influenza immunization is recommended because protection is short-lived and the vaccine composition changes. However, the efficacy and effectiveness of this intervention is largely unproven. Not surprisingly, studies have shown that lung transplant patients have lower antibody responses than healthy individuals do. To this end, this study tests the hypothesis that the influenza vaccine-induced T cell responses will be similar in lung transplant patients and healthy individuals.

Blood will be drawn prior to and 2-4 weeks after immunization and used to measure antibody responses by hemagglutination inhibition assay.

Samples will be collected in Jan-April each season to study Trans-vivo Delayed Type Hypersensitivity (TVDTH) response.

[This substudy that was originally registered to NCT00205270 and subsequently registered to its own NCT number for the purpose of clarity in linked results]

ELIGIBILITY:
Inclusion Criteria:

* Post-lung transplant at University of Wisconsin Hospital
* Healthy adult

Exclusion Criteria:

* Allergy to eggs
* Moderate to severe febrile illness
* Active treatment for acute rejection
* Received season's influenza vaccine prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Post-lung transplant patients at the UW Hospital and healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2004-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Antibody response to influenza vaccine | 2-4 weeks post-immunization (2004-2005 season), up to 1 year (2-4 weeks post-immunization, 2005-2006 season)
  Blood was drawn prior to and 2-4 weeks after immunization and used to measure antibody responses by hemagglutination inhibition assay
T cell response to influenza vaccine antigens | between January and April 2005, between January and April 2006
  T cell response is measured with trans-vivo delayed-type hypersensitivity assay (TVDTH). To induce TVDTH responses, prepared lymphocytes were injected into the footpads of anesthetized (isoflurane) severe combined immunodeficiency (SCID) mice using a 0.5 ml syringe with a 28-gauge needle. The resulting swelling is an index of human T cell sensitization.

CONTACTS AND LOCATIONS:
Overall Officials: Mary S Hayney, PharmD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hayney MS, Moran J, Wiegert NA, Burlingham WJ. Lung transplant patients' T cell responses to influenza vaccine viruses between seasons. Vaccine. 2008 May 19;26(21):2596-600. doi: 10.1016/j.vaccine.2008.03.012. Epub 2008 Mar 31. PMID 18420314